CLINICAL TRIAL: NCT03318250
Title: TransGrade Multimodal Neuromodulation of the Dorsal Root Ganglion Ensemble for Refractory Neuropathic Pain: Clinical Efficacy and Procedural Efficiency
Brief Title: TransGrade Multimodal Neuromodulation of the Dorsal Root Ganglion Ensemble for Refractory Neuropathic Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated early at the request of Sponsors.
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DRAGON17; 228782 (Other: IRAS)
Record Dates: First submitted 2017-10-04; First posted 2017-10-23 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Neuropathic Pain; Pain, Chronic
Keywords: DRG Stimulation
MeSH Terms: conditions — Neuralgia; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Burst3D (Active Comparator): This is a device progamme setting which is being compared against DR6-LF.
  Intervention for this arm is the dorsal root ganglion neurostimulation device implant which will occur at trial implant. Once device is implanted participants are assigned progammes in a randomized manner.
  Interventions: Device: Dorsal Root Ganglion Stimulation
- DRG-LF (Active Comparator): This is a device progamme setting which is being compared against Burst3D.
  Intervention for this arm is the dorsal root ganglion neurostimulation device implant which will occur at trial implant.Once device is implanted participants are assigned progammes in a randomized manner.
  Interventions: Device: Dorsal Root Ganglion Stimulation

INTERVENTIONS:
Device: Dorsal Root Ganglion Stimulation — During the Dorsal Root Ganglion implant , SCS leads will be implanted using a TransGrade Dorsal Root Ganglion Technique. Antibiotic prophylaxis is performed prior to surgery for both trial and permanent implant phase. Using the technique lead placement will be performed through a small skin incision under local anaesthesia supplemented by conscious sedation. The leads will be placed along the DRG to obtain stimulation coverage over as much of the pain area as possible. After the leads have been implanted, x-ray or fluoroscopy images will be taken to record the final lead locations. Once intervention is completed participants will assigned either DRG-LF and Burst3D device programme.

SUMMARY:
This a single center study comparing two forms of electrical stimulation: sub-sensory burst stimulation (DRG-Burst3D) and standard low frequency stimulation (DRG-LF) in the dorsal root ganglion of subjects diagnosed with neuropathic pain

DETAILED DESCRIPTION:
The study will consist of two phases; a 26 day randomized trial phase in which the subject will assess the effectiveness of DRG-Burst3D and DRG-LF, and a 12 month post permanent implant follow up phase.

The randomized trial phase which consists of two phases Trial Assessment 1 and Trial Assessment 2 will last for a maximum of 26 days. Subjects will be randomized 1:1 to receiver 10 ±3 days of DRG-LF stimulation and 10 ±3 days of Burst3D stimulation (DRG-Burst3D) to assess the efficacy of each the different forms of stimulation throughout the trial phase.

Subject will complete in clinic questionnaires (SF-36, ODI, DN4, PGIC, Paraesthesia Map) during the trial phase along with multi-day diary to record VAS pain scores. The subject-reported data from multi day diary and in-clinic assessments will be the basis of verification for success of trial (> 50% overall pain relief). Following device trial subjects will take a questionnaire on program preferences of DRG-LF or Burst3D.

If VAS score during either of the two trial assessments is reduced by at least 50% compared to the baseline score, the subject will be considered for permanent DRG-SCS implant. Subjects who do not experience a >50% overall pain relief on either of the two stimulation settings will exit the study.

Subject who underwent a successful trial (> 50% overall pain relief) will then be implanted with Boston scientific Precision NoviTM neurostimulator trial System. Post permanent implant subjects will receive both DRG-LF and Burst3D programs and use their preferred stimulation program.

The subjects will then be followed for 12 months to assess the long-term treatment outcome. Follow up visits will occur at 1, 3, 6 and 12 months after permanent implant. During each of these visits subjects will rate their pain using the VAS, their quality of life using the EQ-5D, their disability using the ODI, Neuropathic pain using DN4 , Mental health using SF-36 and sensation using paraesthesia Map.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old at the time of informed consent
2. Subject is willing and able to provide a signed and dated informed consent
3. Subject is capable of independently comprehending and consenting to the requirements of the study
4. Subject is willing and able to comply with all study procedures, study visits, and be available for the duration of the study
5. Subject has been diagnosed with Neuropathic Pain with VAS pain scores ≥ 6 for at least 6 consecutive months
6. Pain distribution localized predominantly to 1 or 2 body dermatomes
7. Subject is on a stable dose (no new, discontinued or changes) of all prescribed pain medications for at least 4 weeks prior to screening and willing to maintain or only decrease the dose of all prescribed pain medications through Trial Assessment 2.
8. Subject has tried appropriate conventional medical management for their pain

Exclusion Criteria:

1. Subject has an active implanted device, whether turned on or off
2. Subject displays current signs of a systemic infection
3. Subject is pregnant or lactating, inadequate birth control, or the possibility of pregnancy during the study
4. Subject has untreated major psychiatric comorbidity
5. Subject has serious drug-related behavioural issues (eg, alcohol dependency, illegal substance abuse)
6. Using greater than 120mg morphine equivalents of opioids daily
7. Structural abnormalities of the spine that may prevent electrode implantation
8. Co-existing disorder of the nervous system that may affect study measurements e.g polyneuropathy
9. Subjects has a requirement for planned MRI scanning in the future
10. Subject is diagnosed with Raynaud disease
11. Subject is diagnosed with Fibromyalgia
12. Subject has any active malignancy or has been diagnosed with cancer and has not been in remission for at least 1 year prior to screening
13. Subject has secondary gains which, in the opinion of the investigator, are likely to interfere with the study
14. Subject is participating or planning to participate in another clinical trial
15. Subject has characteristics/limits of household or close contacts involved in study (eg, family member already a study participant where blind could be broken)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Pain VAS | 12 Months
  To assess improvements in pain

SECONDARY OUTCOMES:
Collection of healthcare utilization data | 12 Months
  To assess operative time, progamming time and the need for reprogamming
Preference Questionnaire | 26 Days
  To assess subject preference between DRG-LF and Burst3D
Douleur Neuropathique 4 questionnaire | 1 Month
  To assess improvements in neuropathic pain
The Short Form 36 Health survey | 12 Months
  To assess improvements in mental health
EuroQol five dimensions questionnaire | 12 Months
  To assess improvements in quality of life
Oswestry Disability index | 12 Months
  To assess changes in disability and health
Patient Global Impression of Change | 12 Months
  To assess patient satisfaction with therapy
Paraesthesia Map | 12 Months
  To assess changes in location of pain sensation and therapy coverage.
Pain Map | Baseline
  To assess location of pain
7 day pain diary | 12 Months
  To assess eligibility and improvements in pain
Patient Satisfaction questionnaire | 12 Months
  To assess Subject satisfaction with therapy

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Al-Kaisy, Principal Investigator — Guy's and St Thomas NHS Foundation Trust
Locations (1):
- Guy's and St Thomas Hospital, London, United Kingdom